CLINICAL TRIAL: NCT00537758
Title: Treatment for Obesity and Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0204015334; R01DK049587 (NIH)
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2007-09

CONDITIONS: Binge Eating Disorder; Obesity
Keywords: binge eating disorder; cognitive behavior therapy; combination therapy; obesity; weight loss; body weight; clinical trial; dietary restriction; overeating; weight control
MeSH Terms: conditions — Binge-Eating Disorder; Obesity; Weight Loss; Body Weight; Hyperphagia | interventions — Cognitive Behavioral Therapy

ARMS (3):
- 1 (Experimental): Cognitive Behavior Therapy
  Interventions: Behavioral: Cognitive Behavior Therapy
- 2 (Experimental): Behavioral Weight Loss Treatment
  Interventions: Behavioral: Behavioral Weight Loss Treatment
- 3 (Experimental): CBT + BWL
  Interventions: Behavioral: CBT and BWL

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy
  Arms: 1
Behavioral: CBT and BWL
  Arms: 3
Behavioral: Behavioral Weight Loss Treatment
  Arms: 2

SUMMARY:
This study is a test of cognitive behavioral therapy(CBT) and behavioral weight loss (BWL) treatments for obese patients with binge eating disorder (BED). The study involves a comparison of three treatment conditions: (1) CBT; (2) BWL, and (3) a sequential (two-part) treatment consisting of CBT followed by BWL.

ELIGIBILITY:
Inclusion Criteria:

* Binge Eating
* Overweight

Exclusion Criteria:

* Pregnancy
* Current cardiac disease
* Serious neurologic illnesses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2002-07

PRIMARY OUTCOMES:
Binge Eating
BMI

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M. Grilo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Psychiatric Research at Congress Place, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Grilo CM, Pittman B. Exploring Dietary Restraint as a Mediator of Behavioral and Cognitive-Behavioral Treatments on Outcomes for Patients With Binge-Eating Disorder With Obesity. Int J Eat Disord. 2024 Dec;57(12):2475-2481. doi: 10.1002/eat.24288. Epub 2024 Sep 9. PMID 39247962